CLINICAL TRIAL: NCT06082492
Title: The Beneficial Value of 18F FDG PET/CT in the Follow-up of Stage III Non-small Cell Lung Cancer Patients: the NVALT31-PET Study
Brief Title: The Beneficial Value of PET/CT in the Follow-up of Stage III Non-small Cell Lung Cancer Patients
Acronym: NVALT31-PET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Amsterdam UMC, location VUmc (Other); Streekziekenhuis Koningin Beatrix (Unknown); Canisius-Wilhelmina Hospital (Other); Diakonessenhuis, Utrecht (Other); Dijklander Ziekenhuis (Other); Deventer Ziekenhuis (Other); Elisabeth-TweeSteden Ziekenhuis (Other); Gelre Hospitals (Other); Groene Hart Ziekenhuis (Other); HagaZiekenhuis (Other); Martini Hospital Groningen (Other); Medisch Spectrum Twente (Other); St. Antonius Hospital (Other); Franciscus &Vlietland (Other); Tjongerschans (Unknown); Maasstadziekenhuis (Unknown); Gelderse Vallei Hospital (Other); Bravis Hospital (Other); Tergooi Hospital (Other); Treant Zorggroep (Unknown); Amphia Hospital (Other); UMC Utrecht (Other); OLVG (Network); Haaglanden Medical Centre (Other); Antoni van Leeuwenhoek Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 114319; NL83288.091.23 (Other: ToetsingOnline)
Record Dates: First submitted 2023-09-27; First posted 2023-10-13 (Actual); Last update posted 2025-02-05 (Actual); Status verified 2024-12

CONDITIONS: Stage III Non-small Cell Lung Cancer
Keywords: 18F FDG PET/CT scans; Follow-up care
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Tomography, X-Ray Computed

STUDY DESIGN:
Intervention Model Description: This is a multicenter randomized controlled clinical trial with a superiority design. At approximately 4 months after the end of curative intent treatment patients will be randomized 1:1 to either the intervention (18F FDG PET/CT) or the control group (usual care, CT-based follow-up). Randomization will be done stratifying for histology and treatment.
  After the start of the study all patients will have regular follow-up visits at 6, 12, 18, 24 months and 36 months after the end of curative intent treatment, as is stated in the Dutch guidelines. In the intervention group these visits will be complemented by a 18F FDG PET/CT scan, while in the control group the visits will only contain a CT scan.
  For patients in the intervention group who give consent for participation in the collection of blood, blood will be drawn around the scan.
  At all time points patients will be asked to fill in the HRQOL and cost-effectiveness questionnaires.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Experimental): The intervention group (n = 345) consists of usual care until 3 years of follow-up (see comparator) with additional whole-body 18F FDG PET/CT scans (from the skull to, at least, the midfemoral region) during follow-up visits at 6 months, 12 months, 18 months, 24 months, and 36 months of follow-up. After the 36-month follow-up period, patients will receive follow-up usual care (i.e. CT-scans).
  The scanning protocol of Boellaard et al (2015) is the basis of all center-specific protocols and therefore will be followed approximately (PET low dose CT 60 minutes post injection with scan trajectory from skull to (at least the) thighs followed by a CT scan).
  Interventions: Diagnostic Test: 18F FDG PET/CT; Diagnostic Test: CT scan
- Control group (care as usual) (Active Comparator): The control group (n = 345) consists of regular follow-up visits with physical check-ups and CT-scans at least every 6 months for the first 2 years and then at least yearly CT-scans until 3 years of follow-up. In case of suspected recurrence/metastasis or inconclusive results of a CT-scan (eg, after radiotherapy), 18F FDG PET/CT should be considered.
  The standard protocol for a diagnostic CT of the thoracic region during IV contrast administration according to the lung tumor protocol will be followed
  Interventions: Diagnostic Test: CT scan

INTERVENTIONS:
Diagnostic Test: 18F FDG PET/CT — Additional 18F FDG PET/CT scans during follow-up visits at 6, 12, 18, 24 and 36 months of follow-up.
  Other Names: Whole body PET/CT scan
  Arms: Intervention group
Diagnostic Test: CT scan — CT of the thoracic region during follow-up visits at 6, 12, 18, 24 and 36 months of follow-up.

SUMMARY:
The primary objective of this study is to compare the 3-year overall survival of stage III NSCLC patients during follow-up surveillance with 18F-Fluorodeoxyglucose Positron Emission Tomography/ Computerized Tomography (18F FDG PET/CT) versus follow-up with conventional CT surveillance.

Participants will receive usual care until 3 years of follow-up (control group) with additional whole-body 18F FDG PET/CT scans during follow-up visits at 6 months, 12 months, 18 months, 24 months, and 36 months of follow-up in the intervention group.

Other tasks include:

* filling in quality of life (QOL) questionnaires at every time point;
* participating in an interview evaluating the addition of the 18F FDG PET/CT scans (optional);
* collecting blood at the follow-up time points for our secondary endpoint (optional).

Researchers will compare the usual care control group with the intervention group to see if the additional 18F FDG PET/CT scans are (cost-)effective.

DETAILED DESCRIPTION:
Stage III non-small cell lung cancer (NSCLC) patients are at high risk of developing recurrences (50-78%) during follow-up. With more effective treatments available for patients with oligometastatic disease, early detection of tumor recurrence can prolong survival and health-related quality of life and thereby lower the disease burden. With the use of 18F FDG PET/CT during follow-up, recurrences may be detected earlier at an oligometastatic state when curative-intent treatment is still possible.

Primary objective:

- The primary objective of this study is to compare the 3-year overall survival of stage III NSCLC patients during follow-up surveillance with 18F FDG PET/CT versus follow-up with conventional CT surveillance.

The secondary objectives of this study are:

* To compare the 2-year overall survival of stage III NSCLC patients during follow-up surveillance with 18F FDG PET/CT versus follow-up with conventional CT-based surveillance (interim analysis);
* To compare the number of detected (symptomatic and asymptomatic) recurrences of stage III NSCLC patients during follow-up surveillance with 18F FDG PET/CT versus follow-up with conventional CT-based surveillance;
* To compare the event-free survival of stage III NSCLC patients during follow-up surveillance with 18F FDG PET/CT versus follow-up with conventional CT-based surveillance;
* To determine the cost-effectiveness of 18F FDG PET/CT versus conventional CT-based surveillance during follow-up of stage III NSCLC patients;
* To compare the effect of 18F FDG PET/CT versus conventional CT-based surveillance on health-related quality of life during follow-up of stage III NSCLC patients;
* To assess the beneficial value of ctDNA in the detection of recurrences during follow-up in stage III NSCLC patients;
* To identify patients' experiences with the additional 18F FDG PET/CT scans in the follow-up of stage III NSCLC patients.
* To assess differences in type of treatment following recurrence during follow-up in stage III NSCLC patients.

Primary analyses will be performed on an intention-to-treat basis as well as per protocol. Kaplan-Meier curves with stratified log-rank 2-sided tests will be used to compare the survival between groups. In case of empty strata, strata will be collapsed. The clinical relevance of the difference will be primarily expressed in terms of 3-year survival of the intervention versus the control group.

ELIGIBILITY:
Eligible for this study are patients with stage III NSCLC (8th edition TNM Classification) who (are about to) start(ed) follow-up care (which may include adjuvant treatment) at a participating hospital. Patients may already be included during their curative intent treatment. Patients enter a screening period that runs until their randomization.

Inclusion Criteria:

To be eligible to participate in this study, a subject must meet all of the following criteria at the timing of randomization:

* Cytological or histologically proven stage III non-small cell lung cancer before start of curative intent treatment
* Treated with curative intent and started follow-up care
* All adjuvant treatments are permitted as co-intervention during follow-up care
* Age 18 years or older
* ECOG Performance Status classification 0-2 at moment of inclusion
* Written and signed informed consent by the patient or patient's representative (with the understanding that consent may be withdrawn by the patient or patient's representative at any time without consequences to future medical care)

Exclusion Criteria:

A potential subject who meets any of the following criteria will be excluded from participation in this study:

* Life expectancy shorter than 6 months at the end of curative intent treatment
* Evidence of recurrence after end of curative intent treatment and before randomization (4 months follow-up)
* Any condition that, in the opinion of the investigator, would interfere with evaluation of the intervention or interpretation of HRQOL or other study results.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 690 (Estimated)
Dates: Start 2024-03-19 (Actual); Primary Completion 2029-04 (Estimated); Study Completion 2029-06 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 3 years after end of curative intent treatment
  Overall survival (OS) will be defined as time from end of curative intent treatment until death or loss to follow-up or end of study defined as 3 years after end of curative treatment.

SECONDARY OUTCOMES:
Number of detected symptomatic and asymptomatic recurrences | Up to 3 years after end of curative intent treatment
  As seen on a scan and/or confirmed by biopsy
Event-free survival (EFS) | 3 years after end of curative intent treatment
  Event-free survival will be defined as time from end of curative intent treatment until a recurrence (disease progression or relapse) or death or loss to follow-up, whichever comes first.
Quality-adjusted life-years ((QALY's) for the cost-effectiveness analysis (CEA)) | Up to 3 years after end of curative intent treatment
  The European Quality of Life Five Dimension Five Level (EQ-5D-5L) will be used to measure quality-adjusted life-years. The scores will be transformed into health utilities using the Dutch tariff. QALY's will be estimated using the area under the curve method.
Hospital and medical resource use (for the CEA) | Up to 3 years after end of curative intent treatment
  Hospital resource use will be taken from the hospital records, and will include all diagnostic testing, treatment information, hospital visits, telephone and email consultations, and medication use. Other medical resource use as measured using an adapted version of the iMTA Medical Consumption Questionnaire (iMCQ) will provide information on visits to the GP or use of paramedical care. The prices associated with resource use will be derived from the Dutch guideline for costing, and tariffs and prices published by the Dutch Health authority. Total costs will be calculated by multiplying resource use by integral cost prices.
Productivity losses (for the CEA) | Up to 3 years after end of curative intent treatment
  The iMTA Productivity Costs Questionnaire (iPCQ) will provide information on productivity losses. Productivity losses will be values by the friction cost method.
Health-related quality of life (HRQOL) | Up to 3 years after end of curative intent treatment collected around the follow-up scans.
  As measured by the European Organization for Research and Treatment of Cancer Core Quality of Life Questionnaire (EORTC-QLQ-C30) and lung module (EORTC-QLQ-LC13). The main HRQOL endpoints are physical functioning and the QLQ-C30 summary score. The QLQ-C30 summary score is calculated as the mean of the combined domains of the QLQ-C30 scale scores (excluding financial impact and a two-item global quality of life scale. All scale score are linearly transformed to 0-100, following EORTC guidelines. Effects on HRQOL will be investigated including all patients with at least one completed follow-up HRQOL questionnaire.
Patients' evaluation of the 18F FDG PET/CT scans | Up to 3 years after end of curative intent treatment collected around the follow-up scans.
  The impact of the additional 18F FDG PET/CT scans in follow-up care on distress will be evaluated using the 6-item Cancer Worry Scale (CWS) and the Hospital Anxiety and Depression Scale (HADS). Moreover, semi-structured interviews with a selection of patients in the intervention group will be conducted (optional).
Blood samples | Up to 3 years after end of curative intent treatment collected around the follow-up scans.
  Blood will be collected of intervention group patients in centers participating in the blood sample collection. For this, three cell-stabilizing tubes will be collected concurrently with the 18F FDG PET/CT scan, when the IV is inserted or at a planned blood test. The tubes will subsequently be sent to the sponsor within 24 hours, where the cell-stabilizing tubes will be centrifuged at room temperature for 10 min at 1600 g. Cell-free plasma will be stored in 5 mL aliquots at -80 °C until DNA isolation. Cell-free DNA will be isolated from 1 ml plasma for mutation analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Iris Walraven, PhD., Principal Investigator — Radboud University Medical Center; Annemarie Becker-Commissaris, PhD./MD., Principal Investigator — Amsterdam UMC
Locations (27):
- Netherlands (27):
  - Tergooi MC, Hilversum, Utrecht
  - Amsterdam UMC, Amsterdam
  - Antoni van Leeuwenhoek/Nederlands Kanker Instituut, Amsterdam
  - OLVG, Amsterdam
  - Gelre Ziekenhuizen, Apeldoorn & Zutphen
  - Amphia Ziekenhuis, Breda
  - Deventer Ziekenhuis, Deventer
  - Ziekenhuis Gelderse Vallei, Ede
  - Máxima Medisch Centrum, Eindhoven & Veldhoven
  - Treant, Emmen
  - Medisch Spectrum Twente, Enschede
  - Groene Hart Ziekenhuis, Gouda
  - Martini Ziekenhuis, Groningen
  - Tjongerschans ziekenhuis, Heerenveen
  - Dijklander Ziekenhuis, Hoorn
  - Canisius Wilhelmina Ziekenhuis, Nijmegen
  - Radboudumc, Nijmegen
  - Bravis Ziekenhuis, Roosendaal
  - Maasstad ZIekenhuis, Rotterdam
  - Franciscus Gasthuis & Vlietland, Schiedam
  - Haaglanden Medisch Centrum, The Hague
  - HagaZiekenhuis, The Hague
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg
  - Diakonessenhuis, Utrecht
  - UMC Utrecht, Utrecht
  - St. Antonius Ziekenhuis, Utrecht & Nieuwegein
  - Streekziekenhuis Koningin Beatrix, Winterswijk

IPD SHARING:
Plan to Share IPD: Yes
Final (definitive) versions of data used for analysis will be made findable and shared for reuse and/or verification. Documentation/codebooks necessary for understanding the data will be made findable and shared for reuse and/or verification. Left-over blood samples will be made findable and can be accessed to share for reuse and/or verification.
  Metadata will be published in DANS. Metadata of the blood samples and scans will also be published in BBMRI. Crossreferences between DANS and BBMRI will be included.
  A DOI will be assigned to the whole dataset published in DANS Data Station Life, Health and Medical Sciences.
Supporting Information: Study Protocol, Analytic Code
Time Frame: Data will become available after NVALT31- PET study investigators have performed the analyses needed for this study.
Access Criteria: All data will be available on request. Access to the data will be guarded by the CMO Radboudumc and the NVALT31-PET data access committee (DAC) and may be requested by other researchers from Radboudumc and Amsterdam UMC. Also, the data can be used in collaboration with other groups (abroad).

REFERENCES:
- [Derived] Billingy NE, Verberkt CA, Bahce I, Hassing MJ, Schoorlemmer J, Sarioglu M, Senan S, Aarntzen EHJG, Comans EFI, Kievit W, Teerenstra S, Jacobs C, Keijser A, Heuvel MMVD, Becker-Commissaris A, Walraven I; The NVALT31-PET Consortium. Beneficial value of [18F]FDG PET/CT in the follow-up of patients with stage III non-small cell lung cancer (NVALT31-PET study): study protocol of a multicentre randomised controlled trial. BMJ Open. 2025 Jul 25;15(7):e103745. doi: 10.1136/bmjopen-2025-103745. PMID 40713037
- See also: Study website — https://www.radboudumc.nl/lopende-onderzoeken/nvalt31-pet-longkankeronderzoek